CLINICAL TRIAL: NCT00490295
Title: Biomarkers for the Detection of Brain Ischemia in Neonates With Congenial Heart Disease Requiring Cardiac Surgery
Brief Title: Biomarkers for Detection of Brain Ischemia
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: IRB00002572
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Disorders
Keywords: biomarkers; brain ischemia; neonates; cardiac surgery; congenital heart disease
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Brain Ischemia; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- newborn cardiac surgical study group

SUMMARY:
Brain injury occurs in one-quarter to one-half of congenital heart defect infants during the perioperative period. A blood test using a biomarker to diagnose brain injury would be important.

Postoperative cerebral ischemia may be decreased by inotropic support, ventilation, medical management aimed at increasing oxygen delivery to the brain. Currently there are no FDA approved blood tests to assess brain ischemia in infants undergoing cardiac surgery.

Specific Aim 1: We will prospectively study 10 neonates (< 30 days of age) undergoing cardiac surgery utilizing cardiopulmonary bypass for arterial switch operation or Norwood operation to determine the specificity and sensitivity of a blood test for brain injury. This aim will be accomplished by analyzing blood samples for S-100 and NSE drawn prior to surgery, once each day following cardiac surgery as long as the patient remains in the intensive care unit (maximum 5 days)and at the time of postoperative brain magnetic resonance imaging. The S-100B and NSE values will then be correlated with brain magnetic resonance imaging studies before cardiac surgery and at following cardiac surgery.

Hypothesis: We expect the concentration of S-100B and NSE will be significantly higher in the blood of neonates with congenital heart disease who have documented brain injury on brain magnetic resonance imaging (MRI). Furthermore, we predict that the blood levels of S-100B and NSE may correlate to clinical outcome (time to extubation, hospital discharge, neurodevelopmental outcome at 6 months of age).

Specific Aim 2: We will prospectively study these neonates at 6 months following cardiac surgery to determine a correlation between neurodevelopment and concentration of S-100B and NSE. To achieve this specific aim, a blood sample for S-100B and NSE and neurodevelopmental testing will be done at 6 months following cardiac surgery.

Hypothesis: We expect neonates with elevated S-100B and NSE and abnormal brain magnetic resonance imaging documented in specific aim 1 to have a significant decline in neurodevelopment at 6 months after cardiac surgery.

Long-term: The long-term goal of this research is to diagnose brain ischemia in infants using a biomarker blood test.

DETAILED DESCRIPTION:
1. Ten full-term neonates (> 36 week gestation), between 1-30 days of age, who present for arterial switch operation or Norwood operation will have 2 ml of blood drawn prior to cardiac surgery, 2 ml blood drawn each day after cardiac surgery as long as the patient remains in the intensive care unit with indwelling lines (maximum of 5 days) and 2 ml blood drawn on the day of the followup brain magnetic resonance imaging study (if not within the maximum of 5 days) to determine blood concentrations S100B and NSE.
2. Brain magnetic resonance imaging (MRI) including T1, 2, DWI, spectroscopy, and magnetic resonance angiography, will be performed prior to cardiac surgery and following cardiac surgery in all study patients. Timing of the follow-up brain magnetic resonance imaging including T1, 2, DWI, spectroscopy, and magnetic resonance angiography, will be based on stability of the patient as assessed by the attending physician. Optimal timing for brain magnetic resonance imaging is 4 days postop.
3. Maternal information including level of education, medications, and medical history will be obtained. Two mls of blood will also be obtained from the mother to determine maternal blood concentrations of S100B and NSE.
4. Study patient clinical variables, including vital signs (heart rate, blood pressure, respiratory rate), systemic oxygen saturation by extremity pulse oximetry, near infrared spectroscopy (NIRS), routine laboratory values will be obtained at the time of each study blood sample.
5. Operative variables including cardiopulmonary bypass time, aortic cross clamp time, circulatory arrest time, and hematocrit on bypass will be obtained. Transfusion quantity of packed red blood cells, fresh frozen plasma, platelets, and cryoprecipitate used in the operating room and in the cardiac intensive care unit will also be obtained
6. Outcome variables including length of mechanical ventilation, hospital stay, and gross neurological abnormalities (clinical seizures) will be obtained.

   Follow-up:
7. All patients will have neurodevelopmental testing at 6 months after heart surgery.
8. Another 2 mls of blood S100B and NSE will be obtained when the patient returns at 6 months for neurodevelopmental testing.

ELIGIBILITY:
Inclusion Criteria:

* Ten consecutive full-term (>36 week gestation) neonates, one day to 30 days of age, presenting for cardiac surgery for arterial switch operation or Norwood operation will be eligible for the study.
* No patient will be excluded because of race or ethnicity.
* Parental or legal guardian consent will be obtained for all patients prior to enrollment.

Exclusion Criteria:

* Newborns with multiple organ abnormalities in addition to their heart defect such as diaphragmatic hernia, tracheo-esophageal fistula, and congenital syndromes involving multiple organs will be excluded from participation.
* Newborns with genetic syndromes associated with developmental delay will also be excluded.
* Newborns with birth asphyxia, 5 minute Apgar score < 5, will be excluded. Patients with multiple organ failure, syndromes, and birth asphyxia have other causes for neurodevelopmental abnormalities.
* Those patients unable to return for postop follow-up and neurodevelopmental testing will be excluded from participation.
* Those patients with parents/guardians who are unable to read or speak English will be excluded from participation.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ten consecutive full-term (>36 week gestation) neonates, one day to 30 days of age, presenting for cardiac surgery for arterial switch operation or Norwood operation will be eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Diagnose brain ischemia in infants using a biomarker blood test. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Simsic, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States